CLINICAL TRIAL: NCT05906615
Title: Intravenous Lidocaine for Pain Associated With Pancreatic Cancer and Chronic Pancreatitis (LIDOPAN)
Brief Title: Intravenous Lidocaine for Pain Associated With Pancreatic Cancer and Chronic Pancreatitis
Acronym: LIDOPAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, M.G. Besselink, prof. M.G. Besselink, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W21_005 # 21.007
Record Dates: First submitted 2022-08-29; First posted 2023-06-18 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Cancer; Chronic Pancreatitis
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenous lidocaine (Other): Monitored intravenous lidocaine infusion for patients with CP and pancreatic cancer is already current practice in the participating centers. Patients undergo treatment in the recovery unit of the anesthesiology department, for early detection of possible, although highly unlikely adverse events such as anaphylactic reactions, arrhythmias or hypotension. At the recovery unit continuous monitoring is possible and treatment of the above mentioned side effects can be easily provided. Continuous monitoring includes a 3-lead ECG, saturation, and blood pressure control every 15 minutes.
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Lidocaine IV — Administration of IV lidocaine will take place according to the standard protocol as is currently already used in daily clinical practice. First, a lidocaine bolus of 1.5mg/kg is administered, followed by a continuous infusion of 1.5mg/kg/hour. When no pain relief is noticed, each 15 minutes the dose is raised with 1ml up to a maximum of 2mg/kg/hour. If again no pain relief is noticed, the anesthesiologist is consulted. When the anesthesiologist agrees, and no side effects occur, lidocaine infusion can be increased up to a maximum of 2.5mg/kg/hour, with a maximum of 250mg/hour. When there is a pain response - pain is reduced with at least two NRS points or 30% from baseline - that dose is administered for two hours continuously. Following treatment the patient will be observed for an hour before leaving the hospital or recovery unit, again, all according to current daily clinical practice.

SUMMARY:
Pain is a major clinical problem for many patients with pancreatic cancer and chronic pancreatitis (CP).In pancreatic cancer, nearly 75% of patients suffer from pain at the time of diagnosis, with over 90% of patients in advanced stages. In CP, pain occurs in 80-90% of patients and strongly affects quality of life. For both conditions, the majority of pain is addressed using the WHO analgesic ladder. However, more invasive pain therapies are often necessary.

Currently, in several centers in the Netherlands, treatment with IV lidocaine is already used in clinical practice in patients with pancreatic cancer and CP. Based on practical experience, the majority of patients benefit from this therapy, however, its efficacy in terms of duration of pain relief, decrease in pain scores, increase in patient satisfaction and adverse events is unknown. Therefore, the aim of this study is to investigate the efficacy of monitored single intravenous infusion in patients with pancreatic cancer and CP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* NRS score ≥4 despite previous pain treatment with non-opioid analgesics, opioids or TCAs. Or pain treatment with non-opioid analgesics, opioids or TCAs with adequate effect on pain, but unable to reduce the opioids;
* For CP:

  * Diagnosis of CP based on the M-ANNHEIM diagnostic criteria;17
* For pancreatic cancer:

  * Diagnosis of pancreatic cancer (all stages)
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
  * Life expectancy ≥ 3 months;
* Consensus of surgeon/gastroenterologist and anesthesiologist for suitability for treatment

Exclusion Criteria:

* Patients with contra-indications for intravenous lidocaine i.e. medical history of non-adequate liver function, hypersensitivity to local anesthetics, New York Heart Association Class III or IV cardiac disease or myocardial infarction within the past 12 months, shock, and conduction abnormalities (defined as second and third degree atrioventricular (AV) blocks, or atrial fibrillation);
* Patients who underwent invasive pain therapies: such as endoscopic treatment or surgery for chronic pancreatitis, and splanchnic nerves or coeliac plexus blocks, neurolysis, or PRF for pancreatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Pain score | Directly after treatment
  Assessed by the Brief Pain inventory (scale: 0-10, higher score indicate worse outcome)

SECONDARY OUTCOMES:
Effect of treatment | After two weeks, and one-three-six months
  Assed by the Global Perceived effect (scale: 0-7, higher score indicate better outcome)
Pain score | Directly after treatment, two weeks, and after one-three-six months
  Assessed by the Numeric Rating Scale (scale: 0-10, higher score indicate worse outcome)
Pain score long term | After two weeks, and one-three-six months
  Assessed by the Brief Pain inventory (scale: 0-10, higher score indicate worse outcome)
Quality of life (SF-12) | Baseline, and after one-three-six months
  Assessed by the SF-12 (scale: 0-100: higher scores indicate better quality of life)
Dose of intravenous lidocaine administered | During intervention
  in mg/kg
Number of total performed treatments with intravenous lidocaine per participant | During follow-up (six months)
Numer of participants with minor or major complications | During follow-up (six months)
Dose reduction of opioids | During follow-up (six months)

CONTACTS AND LOCATIONS:
Overall Officials: Marc G. Besselink, MD PhD MSc, Principal Investigator — Amsterdam UMC, Academic Medical Center
Locations (1):
- Amsterdam UMC, locatie AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No